CLINICAL TRIAL: NCT01795599
Title: Cervical Preparation for Surgical Abortion at 12-14 Weeks: a Prospective, Randomized, Evaluator-blinded, Multicenter, Controlled Comparison Between Mifepristone, Misoprostol and Their Combination
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-005276-34; 2012-36 (Other: AP HM)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Surgical Abortion
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- mifepristone/misoprostol (Experimental)
  Interventions: Drug: Mifegyne ®; Drug: Gymiso®
- misoprostol (Active Comparator)
  Interventions: Drug: Gymiso®
- mifepristone (Active Comparator)
  Interventions: Drug: Mifegyne ®

INTERVENTIONS:
Drug: Mifegyne ®
  Arms: mifepristone; mifepristone/misoprostol
Drug: Gymiso®
  Arms: mifepristone/misoprostol; misoprostol

SUMMARY:
More than 100 000 surgical abortions are annually performed in France. About four in ten women will have an abortion in their life. Abortion complications are cervical tearing (0.1-1.18%), uterine perforation (0.09-19.8‰), hemorrhage (1.5‰) and infection (5-20%). These complications can first compromise the vital prognosis and are involved in 10% of the worldwide maternal mortality (20 000 women by year), then lead to infertility which is hard to treat (uterine synechiae) or impossible to treat (hysterectomy for control of bleeding), and are finally responsible for obstetrical pathologies as late miscarriages or premature delivery due to cervical insufficiency. All that complications are linked to cervical laceration of the surgical abortion, that can be reduced by the recommended use of mifepristone or misoprostol as cervical preparation for the abortions after 12 weeks. However, it does not exist data evaluating the superiority of one of the two molecules or their combination. These data could optimize the cervical preparation and thus reduce the abortion complications with a direct impact on maternal mortality, infertility and obstetrical complications. Thus, it seems to be important to evaluate these two molecules and their combination.

Objectives To compare mifepristone, misoprostol and their combination in the cervical preparation of the surgical abortion between 12 and14 weeks for their efficacy, complications and side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Woman of 18 or more years old;
* Woman presenting a only intra-uterine pregnancy, the term of which is upper to 11 LIMITED COMPANIES 6 days and inferior strictly to 14 LIMITED COMPANIES, estimated(esteemed) by echography by a measure of the crânio-caudal length included between 55 and 84 millimeters; ·Woman wishing a TERMINATION OF PREGNANCY;

Exclusion Criteria:

* minor Woman;
* Woman presenting a multiple pregnancy;
* Woman presenting an uterine deformation (compartmentalized womb, cocked hat, fibroid praevia);
* Woman presenting a disorder of the coagulation defined by biological parameters (TP(BUSINESS RATE,PRACTICAL CLASS,PRACTICAL CLASSES) < 70 %, TCA report(relationship) patient / witness < 1,20);
* Woman presenting an allergy or a sentimentality known about one of the active substances or about one of the excipients;
* Woman presenting a contraindication to the mifepristone: chronic suprarenal insufficiency, unchecked severe asthma by treatment(processing), porphyrie hereditary, allergy was known about the active substance or about one of the excipients;
* Woman presenting a contraindication to the misoprostol: sentimentality in the active substance, in one of the excipients or in the other prostaglandines;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
reduction of the bleeding | 24month

SECONDARY OUTCOMES:
reduction of the complications | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France